CLINICAL TRIAL: NCT05467202
Title: To Evaluate the Safety and Efficacy of CLL1 CAR-T in Patients With Relapsed and Refractory Acute Myeloid Leukemia
Brief Title: Evaluate the Safety and Efficacy of CLL1 CAR-T in Patients With R/R AML
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, He Huang, Professor, Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BG-CT-22-002(CLL1)
Record Dates: First submitted 2022-07-01; First posted 2022-07-20 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: AML

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group (Experimental): Dose Escalation:After enrollment ,Participants complete the PBMC apheresis,then complete the Lymphocyte clearance,and then receive the dose climning test: 3×10e6/kg，6 ×10e6/kg，9×10e6/kg.
  Dose Expansion:Participants receive a single dose (at the MTD determined).
  Interventions: Drug: CLL1 CAR-T

INTERVENTIONS:
Drug: CLL1 CAR-T — A single infusion of autologous CLL1 CAR-T cells administered intravenously

SUMMARY:
This is an open label, phase I study to assess the safety and efficacy of CLL1 CAR-T in patients with relapsed and refractory acute myeloid leukemia

ELIGIBILITY:
Inclusion Criteria:

1. All subjects must sign and date the Informed Consent before initiating any study specific procedures or activities;
2. Diagnosed as relapse/refractory (r/r) de novo or secondary acute myeloid leukemia (AML);
3. The expression of CLL1 in AML blast is positive ;
4. The patient has recovered from the toxicity of previous treatment;
5. ECOG score ≤ 2 and expected survival period is not less than 3 months;
6. Adequate organ function defined as:

   AST ≤3×ULN; ALT ≤3×ULN; Total bilirubin ≤1.5×ULN; Serum creatinine ≤1.5×ULN, or CCR≥60 mL/min; Hemoglobin ≥60g/L ; Indoor oxygen saturation ≥92%; LVEF≥45%;
7. Pregnancy testing: females of childbearing potential must have a negative serum or urine pregnancy test;
8. From the use of study drug to 2 years after treatment, males and female of childbearing potential must agree to use an effective method of contraception

Exclusion Criteria:

1. Diagnosis of acute promyelocytic leukemia;
2. History or presence of a CNS disorder;
3. HBsAg or HBcAb are positive; HCV 、HIV and Syphilis antibody are positive, CMV DNA in peripheral blood is more than≥500 copies /mL;
4. History of severe hypersensitivity reaction;
5. History of myocardial infarction, cardiac angioplasty or stenting, unstable angina, New York Heart Association Class II or greater congestive heart failure, atrial fibrillation, or other clinically significant cardiac disease within 12 months before enrollment;
6. History of organ transplant surgery;
7. Required systemic application of immunosuppressive or other drugs;
8. Auto-SCT within the 3 months before enrollment;
9. Active autoimmune or inflammatory diseases of the nervous system (e.g., Guillain-Barre syndrome (GBS), amyotrophic lateral sclerosis (ALS)) and clinically active cerebrovascular diseases (e.g., cerebral edema, posterior reversible encephalopathy syndrome (PRES));
10. Requirement for urgent therapy due to ongoing or impending oncologic emergency (eg, leukostasis or tumor lysis syndrome (TLS)) ;
11. Presence or suspicion of a fungal, bacterial, viral, or other infection that is uncontrolled or requiring antimicrobials for management;
12. Live vaccine received within the ≤ 4 weeks before enrollment;
13. Persons with serious mental illness;
14. History of major surgical operations four weeks before enrollment;
15. History of alcoholism or substance abuse;
16. Was identified by the investigators as unsuitable to participate in the study

Ages: 2 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-08-01 (Estimated); Primary Completion 2024-08-02 (Estimated); Study Completion 2025-08-02 (Estimated)

PRIMARY OUTCOMES:
Evaluation of Safety | Up to 2 years after CLL1 CAR-T infusion
  Count the Incidence of adverse events
Changes in cytokine level after CLL1 CAR-T infusion | Up to 2 years after CLL1 CAR-T infusion
  Calculate the change of cytokine level in peripheral blood by flow cytometry after CLL1 CAR-T infusion. Cytokines include IL-2、IL-6、IL-10、IFN-γ.

SECONDARY OUTCOMES:
Complete response rate(CRR) | Up to 2 years after CLL1 CAR-T infusion
  Proportion of subjects who achieved morphological complete response (CR) and complete response with hematologic incomplete recovery (CRi)
Partial response Rate (PRR) | Up to 2 years after CLL1 CAR-T infusion
  Proportion of subjects who achieved a partial response (PR)
Overall response Rate(ORR) | Up to 2 years after CLL1 CAR-T infusion
  Proportion of subjects who achieved CR, CRi, or PR

OTHER OUTCOMES:
Overall survival | Up to 2 years after CLL1 CAR-T infusion
  Death from any cause from the beginning of cell transfusion
Recurrence free survival (RFS) | Up to 2 years after CLL1 CAR-T infusion
  From remission to relapse or death of the subject (including all causes), whether the subject relapsed or died is unknown until the date of the last follow-up examination.
Event-free survival (EFS) | Up to 2 years after CLL1 CAR-T infusion
  Counting from the beginning of cell transfusion until treatment failure, recurrence, or death (various causes). Subjects without any of these events were counted up to the last follow-up examination date. For patients without CR or CRi, EFS is calculated from the beginning of cell transfusion until disease progression or death. Based on the initial event.
MRD negative rate | Up to 2 years after CLL1 CAR-T infusion
  The rate of MRD negative subjects was determined by flow cytometry.
Median BM Reduction | Up to 2 years after CLL1 CAR-T infusion
  Changes of bone marrow primitive cells after cell transfusion from baseline.
Percentage of subjects disengaged from transfusion | Up to 2 years after CLL1 CAR-T infusion
  Percentage of baseline transfusion-dependent subjects who were discharged from transfusion after cell transfusion.

CONTACTS AND LOCATIONS:
Overall Officials: He Huang, MD, Principal Investigator — The First Affiliated Hospital, Zhejiang University
Locations (1):
- The First Affiliated Hospital, Zhejiang University, Hangzhou, China